CLINICAL TRIAL: NCT06509620
Title: Physical and Cognitive Performance in Older Adults With Fatigue
Status: Not yet recruiting | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Doha Rasheedy, Professor of Geriatrics and Gerontology, Ain Shams University
Other Study IDs: MS313/2024
Record Dates: First submitted 2024-07-10; First posted 2024-07-19 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: Fatigue
Keywords: fatigue; older adult
MeSH Terms: conditions — Fatigue | interventions — Mental Status and Dementia Tests

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- cases: community dwelling elderly patients with fatigue. 70 Participants aged 60 years old and above both males and females with fatigue for at least 4 weeks not due to acute condition
  Interventions: Other: Fatigue severity scale
- control: age and gender matched elderly patients without fatigue
  Interventions: Other: Fatigue severity scale

INTERVENTIONS:
Other: Fatigue severity scale — fatigue severity scale is a unidimensional, nine-item questionnaire capturing information on the impact and severity of fatigue. Participants rated the 9-items on a 7-point, Likert-type scale with anchors of strongly disagree (1) and strongly agree (7) based on the previous week. The overall score is an average of the individual item scores and can range between 1 and 7.
  Other Names: Modified Fatigue Impact Scale; MONTREAL COGNITIVE ASSESSMENT; 6 Minute walk test

SUMMARY:
Fatigue is a common symptom in older adults, often linked to various medical conditions, medications, and psychosocial factors, and it can adversely affect both physical and cognitive performance in the aging population, contributing to functional decline and reduced quality of life.

Assessment of the physical impact of fatigue on physical and cognitive performance in older adults can offer valuable insights for clinical practice and holistic geriatric care. Therefore, this study will validate subjective tools used for measuring the impact of fatigue against objective measures.

ELIGIBILITY:
Inclusion Criteria:

* Participants aged 60 years old and above both males and females

Exclusion Criteria:

* o Patients with acute medical illness.

  * Patients with life threatening illnesses.
  * Bedridden patients.
  * Patients with diagnosed malignancy.
  * Patients with debilitating chronic disease (end organ failure) (e.g. heart failure , renal failure, and liver cell failure).
  * Patients with neurological diseases (e.g. moderate to severe dementia, stroke, parkinsonism) that interfere with the assessment process.
  * Patients with musculoskeletal conditions that interfere with the assessment process (fracture, disabling osteoarthritis, painful arthritis).
  * Patients with severe uncorrected hearing loss, vision impairment, or aphasia that may impede effective communication during the assessment.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Community dwelling elderly participants (caregivers of inpatients, attendants of primary care , elderly clubs and other community gatherings).
Sampling Method: Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
The primary outcome measure the difference in cognitive performance between older adults with and without fatigue, assessed using the Montreal Cognitive Assessment (MoCA) | 6 months
  compare the MoCA scores between the fatigued and non-fatigued groups using appropriate statistical methods (e.g., t-tests or ANCOVA adjusting for potential confounders). MOCA score is 30 with 18-25 = mild cognitive impairment, - 10-17= moderate cognitive impairment and - less than 10= severe cognitive impairment.
The primary outcome measure the difference in physical performance between older individuals with and without fatigue, assessed using 6 minutes walk test | 6 months
  The primary outcome will compare the 6 minutes walk test between the fatigued and non-fatigued groups using appropriate statistical methods (e.g., t-tests or ANCOVA adjusting for potential confounders).

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided